CLINICAL TRIAL: NCT01510834
Title: Computerized Tailored Intervention for Behavioral Sequelae of Post-Traumatic Stress Disorder in Veterans
Brief Title: Computerized Tailored Intervention for Behavioral Sequelae of PTSD in Veterans
Acronym: CTI-PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pacific Islands Health Care System (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Pro-Change Behavior Systems (Other); University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-04/JLS 0002; W81XWH-09-2-0106 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2011-10-07; First posted 2012-01-18 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2013-07

CONDITIONS: Post Traumatic Stress Disorder; Smoking; Anxiety; Depression
Keywords: Computerized Tailored Intervention; CTI; Post Traumatic Stress Disorder; PTSD; Smoking; Anxiety; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Smoking; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All STR2IVE Participants (Experimental): All participants who met study criteria, consented and were enrolled, were asked to complete online assessments at three timepoints(baseline, 1-month, and 3-months) and complete 2 or more behavioral programs each month. Behavioral programs and assessments were provided online via the Multibehavioral, Computerized Tailored Intervention STR2IVE.
  Interventions: Behavioral: Multibehavioral, Computerized Tailored Intervention STR2IVE

INTERVENTIONS:
Behavioral: Multibehavioral, Computerized Tailored Intervention STR2IVE — All participants were provided with the same multibehavioral CTI system and chose two or three behavior programs to complete (smoking cessation, stress management, and/or depression prevention)monthly. They were asked to complete an assessments at baseline, 30-days, and 90-days. They were allowed to access the system workbook anytime but they must wait a minimum of 25 days between assessments and programs at time points 1 and 2, and 55 days between time points 2 and 3.

SUMMARY:
This project assesses the usability and feasibility of a multi-behavioral computerized, tailored intervention (CTI) or expert system delivered via the Internet for veterans with Post-Traumatic Stress symptoms. Three behavioral health risk factors, (1) smoking, (2) depression, and (3) stress, that are associated with Post-Traumatic Stress Disorder (PTSD), are included in the Computerized, Tailored Intervention (CTI) system. The project adapts and modifies an existing CTI system built on the Transtheoretical Model of Behavior Change (TTM) to make it relevant to a veteran population. The system has been successfully utilized with general adult populations. The study utilizes methods that are characteristic of a product development project. Each of the four project phases are sequential and build upon the results of the previous phase. Phase 1 focuses on the review of current CTI programs on smoking cessation, stress management, and depression prevention, and integrating them into a multi-behavioral program for application with veterans. Phase 2 includes the development and adaptation of text-based feedback messages and multimedia components for smoking cessation, stress management, and depression prevention for veterans. Initial testing of the modified CTI programs commences in Phase 3. Cognitive and usability testing with veterans are performed, and additional modifications to the behavioral modules are made based on the test results. Phase 4 focuses on a feasibility study to test the multi-behavioral CTI system with veterans online.

DETAILED DESCRIPTION:
This proof of concept project develops and pilot tests a viable Internet-based intervention to assist veterans with Post-Traumatic Stress symptoms to progress toward changing negative health behaviors that are associated with PTSD and are often difficult to change. Most commercially available CTIs and software applications have limited impact, because of the lack of theory-driven material and empiricism. The proposed CTI is supported by more than 30 years of scientific evidence, and uses the Transtheoretical Model of Behavior Change (TTM) as the theoretical basis for generating personalized interventions (Prochaska & Velicer, 1997; Velicer, Prochaska, & Redding, 2006). The TTM is ideally suited to those who are resistant to change and unlikely to take action in the near future, as well as those prone to relapse.

The intervention will be primarily targeted at negative coping strategies that confound or exacerbate Post-Traumatic Stress symptoms and hinder progress toward remission. Progress in a Transtheoretical Model of Behavior Change (TTM) conceptual framework may be defined as movement from one TTM stage of change to the next level of the change process, rather than the elimination or significant reduction of smoking, depression, or stress per se. The CTI system that will be modified during this project has been empirically tested and validated with a general population and has demonstrated significant outcomes for the three proposed modules - smoking cessation, depression prevention, and stress management. The CTI system provides an intervention that emphasizes advancement through the processes of change at one's own pace as the focus of project, rather than the linear progression through a structured behavior change program to achieve changes in the undesired behaviors.

Hypothesis 1: The structure and TTM-based content of the adapted Smoking Cessation, Depression Prevention, and Stress Management systems and consequent CTI will be appropriate for veterans.

Primary Aim 1: To modify TTM-based Smoking Cessation, Depression Prevention, and Stress Management behavioral intervention modules, originally developed for general adult populations, to be appropriate and relevant for veterans with Post-Traumatic Stress symptoms.

Secondary Aim 1a: To conceptualize the CTI program's approach, content, and design based on input from a diverse sample of military veterans and expert consultants.

Hypothesis 2: A multi-behavioral CTI can be successfully implemented with veterans who have Post-Traumatic Stress symptoms

Primary Aim 2: To demonstrate that a multi-behavioral CTI can be successfully implemented with veterans with Post-Traumatic Stress symptoms.

Secondary Aim 2a: To conduct usability interviews with veterans to ensure that the target population can navigate through the computerized intervention and understand the intervention content.

Secondary Aim 2b: To demonstrate the feasibility of CTI by: a) recruiting veterans to the project and delivery of the proposed intervention; and b) assessing the acceptability and perceived usefulness of the intervention from the perspective of veterans with Post-Traumatic Stress symptoms.

Secondary Aim 2c: To demonstrate feasibility of CTI to increase motivation to change targeted behaviors, i.e., smoking cessation, depression prevention, and stress management.

Secondary Aim 2d: To demonstrate positive change in assessment outcomes for Post-Traumatic Stress symptoms, depression, quality of life, and perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* Military Veterans, Operation Iraqi Freedom (OIF)/Operation Enduring Freedom (OEF) service preferred
* 18 years or older
* Ability to read and comprehend English
* Mild to moderate PTSD symptoms
* Cigarette smoking (preferred)
* Mild to moderate depression (preferred)
* Difficulty managing stress
* Comfortable using a computer and access to the Internet

Exclusion Criteria:

* Present with psychosis, bipolar disorder, active substance use, or cognitive impairment
* Severe depression or suicidal ideation (Patient Health Questionnaire-9)(PHQ-9 >19)
* Severe PTSD symptoms (PTSD Symptom Checklist)(PCL-M >73)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Spira, Ph.D., Principal Investigator — National Center for PTSD Pacific Islands Division
Locations (3):
- United States (3):
  - VA Pacific Island Health Care System, Honolulu, Hawaii
  - Dept of Public Health, John A. Burns School of Medicine, University of Hawaii at Manoa, Honolulu, Hawaii
  - Pro-Change Behavioral Systems, Inc., Kingston, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordan PJ, Evers KE, Burke KY, King LA, Nigg CR. A computerized, tailored intervention to address behaviors associated with PTSD in veterans: rationale and design of STR(2)IVE. Transl Behav Med. 2011 Dec;1(4):595-603. doi: 10.1007/s13142-011-0088-1. PMID 24073082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from July 22, 2011-November 30, 2011. Recruitment was accomplished through targeted mailings to VA patients at risk for PTSD; study flyers at VA mental health providers; and social media networks to target veterans. Pre-screening, consenting, assessments, enrollment, and intervention were done completely online.
Pre-assignment Details: To minimize participant risk, secondary screening excluded veterans who did not meet risk criteria for mild to moderate PTSD (score <25 or >73 on the PCL-M), or had severe depression (scoring ≥20 on the PHQ-8). 354 veterans registered on the site, 95 did not complete screening; 169 screened out; 90 completed baseline assessments.
Groups:
- All Participants: All participants who met study criteria, consented and were enrolled, were asked to complete online assessments at three timepoints(baseline, 1-month, and 3-months) and complete 2 or more behavioral programs each month.
Period: Overall Study
Arm/Group | All Participants
Started | 90
Completed | 57
Not Completed | 33

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 68
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Change in PCL-M Score (PTSD Symptom Checklist-Military [PCL-M], Weathers et al., 1993)
Description: Developed by researchers at the VA National Center for PTSD, PCL is a self-report questionnaire that consists of 17 questions that map directly onto DSM-IV criteria for PTSD. Respondents are asked how often they have been bothered by each symptom in the past month on a 5-point Likert scale (1=not at all to 5=extremely). Previous research has shown internal consistency coefficients were high for the total scale (.97) and for each subscale (.92 - .93). Test-retest reliability over 2-3 days was shown to be .96. Scores can range from 17-85, with a score of 48 typically indicating PTSD in military populations. The National Center for PTSD recommends using 5 points as a minimum threshold for determining whether an individual has responded to treatment and 10 points as a minimum threshold for determining whether the improvement is clinically meaningful. A higher score indicates more PTSD symptoms, therefore, a score reduction from T1 to T3 is a better outcome than an increase.
Time Frame: Change in PCL-M score from baseline (T1) to final 3 mos. follow-up (T3)
Population: 57 completing all time points for intervention and assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Difference in PCL (T1, T3) (Negative Change is Better): Mean difference in PCL (T1, T3) for study completers
Arm/Group | Mean Difference in PCL (T1, T3) (Negative Change is Better)
Number analyzed (Participants) | 57
units on a scale | -6.82456 (14.1486)
Statistical Analysis 1: Comparison: Mean Difference in PCL (T1, T3) (Negative Change is Better); Test type: Superiority or Other; p = .001, t-test, 2 sided; Mean Difference (Final Values) = -6.824, 95% CI 2-sided [-10.578 to -3.070], Standard Deviation 14.148

2. Secondary Outcome: Change in QOLS Score T1 to T3 (Quality of Life Scale [QOLS], Flanagan, 1978, 1982)
Description: The QOLS contains 16 items that represent five conceptual domains of quality of life. QOLS was developed with more consideration to cultural diversity and individual perspectives than other commonly used measures. It uses a unique 7-item Likert scale that allows responses regarding different aspects of life to range from "delightful" to "terrible". It has been found to be internally consistent with alpha from .82 to .92 and showed high test-retest reliability over 3-weeks (r = 0.78 to r = 0 .84). The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112. Previous validation research showed that patients who participated in a treatment program and rated their symptoms as improved by 60% or gained on average 7 to 8 points on the QOLS total score. A higher QOLS score indicates better quality of life, therefore, a positive score change is a better outcome.
Time Frame: Change in QOLS score from baseline (T1) to final 3 mos. follow-up (T3)
Population: Participants completing all 3 study time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Difference in QOLS (T1, T3): Mean Difference in QOLS (T1, T3)for study completers only
Arm/Group | Mean Difference in QOLS (T1, T3)
Number analyzed (Participants) | 57
units on a scale | 7.08772 (15.73132)
Statistical Analysis 1: Comparison: Mean Difference in QOLS (T1, T3); Test type: Superiority or Other; p = .001, t-test, 2 sided; Mean Difference (Final Values) = 7.0872, 95% CI 2-sided [2.91 to 11.26], Standard Deviation 15.731

3. Secondary Outcome: Change in PSS From T1 to T3 (The Perceived Stress Scale [PSS] Cohen, Kamarck, & Mermelstein, 1983)
Description: The PSS is the most widely used psychological instrument for measuring the perception of stress. It is a 10-item questionnaire that measures an individual's subjective evaluation the stressfulness of situations in their life in the past month. Items are designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The items are of a general nature and relatively free of content specific to any subpopulation. Internal consistency reliability of the PSS has been shown to be moderate (Cronbach alpha coefficient =.78) and that it has good test-re-test reliability. Scores can range from 0-40 as items are scored 0-4 points each. A higher score indicates more stress, so a negative change from baseline (T1)to 3-month follow-up (T3) is a better outcome.
Time Frame: Change in PSS score from baseline (T1) to final 3 mos. follow-up (T3)
Population: All participants completing all 3 time points of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Difference in PSS (T1, T3): Mean difference in Perceived Stress Scale (T1, T3) for study completers
Arm/Group | Mean Difference in PSS (T1, T3)
Number analyzed (Participants) | 57
units on a scale | -3.78 (7.79)
Statistical Analysis 1: Comparison: Mean Difference in PSS (T1, T3); Test type: Superiority or Other; p < .001, t-test, 2 sided; Mean Difference (Final Values) = -3.78, 95% CI 2-sided [-5.84 to -1.70], Standard Deviation 7.78

4. Secondary Outcome: Change in PHQ-8 From T1-T3 (Patient Health Questionnaire [PHQ-8], Kroenke & Spitzer, 2002; Spitzer, Kroenke, & Williams, 1999)
Description: The PHQ-9 is the self-administered depression module of the Patient Health Questionnaire that assesses common mental disorders. Eight of the 9 items in the scale are included in the Depression Prevention Assessment and is also known as the PHQ-8. Item 9, which assesses suicidality has been omitted in the online version. The PHQ-8 has been shown to have a sensitivity of 81% and specificity of 99% for scores 15 and above in diagnosing major depression, with a positive predictive value of 94%. Scores range from 0 to 24 (0-3 points per question multiplied by 8 questions), with 0-9 indicating no depression, 10-14 minor depression, 15-19 moderately severe major depression, and >19 indicating sever major depression. An initial drop of 5 points is considered adequate treatment response for 3 counseling sessions over 4-6 weeks. A higher score indicates more depression, so a reduction in score from baseline (T1) to 3-month follow-up (T3) is a better outcome.
Time Frame: Change in PHQ-8 score from baseline (T1) to final 3 mos. follow-up (T3)
Population: Those participants who completed all 3 time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Difference in PHQ-8 (T1, T3): Mean Difference in PHQ-8 (T1,T3) for study completers
Arm/Group | Mean Difference in PHQ-8 (T1, T3)
Number analyzed (Participants) | 57
units on a scale | -2.08772 (6.26863)
Statistical Analysis 1: Comparison: Mean Difference in PHQ-8 (T1, T3); Test type: Superiority or Other; p = .015, t-test, 2 sided; Mean Difference (Final Values) = -2.08, 95% CI 2-sided [-3.751 to -.4244], Standard Deviation 6.269

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No